CLINICAL TRIAL: NCT03922633
Title: A Phase 1 Clinical Study of a Single Intravenous Dose of E3112 in Japanese Healthy Adult Male Subjects
Brief Title: A Single Intravenous Dose of E3112 in Japanese Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E3112-CP2
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2020-03

CONDITIONS: Healthy Male Participants
Keywords: E3112; Phase 1; Pharmacokinetics; Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 Group A: E3112 + Placebo (Experimental): E3112 intravenous infusion in treatment stage 1 followed by placebo intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 1 Group B: Placebo + E3112 (Experimental): Placebo intravenous infusion in treatment stage 1 followed by E3112 intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 2 Group A: E3112 + Placebo (Experimental): E3112 intravenous infusion in treatment stage 1 followed by placebo intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 2 Group B: Placebo + E3112 (Experimental): Placebo intravenous infusion in treatment stage 1 followed by E3112 intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 3 Group A: E3112 + Placebo (Experimental): E3112 intravenous infusion in treatment stage 1 followed by placebo intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 3 Group B: Placebo + E3112 (Experimental): Placebo intravenous infusion in treatment stage 1 followed by E3112 intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 4 Group A: E3112 + Placebo (Experimental): E3112 intravenous infusion in treatment stage 1 followed by placebo intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo
- Cohort 4 Group B: Placebo + E3112 (Experimental): Placebo intravenous infusion in treatment stage 1 followed by E3112 intravenous infusion in treatment stage 2. A washout period of 7 days will be maintained between the two treatment stages.
  Interventions: Drug: E3112; Other: Placebo

INTERVENTIONS:
Drug: E3112 — Intravenous infusion.
Other: Placebo — Intravenous infusion.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics after a single intravenous dose of E3112 in Japanese healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking Japanese males aged 20 to 44 years at the time of written, informed consent
2. Body Mass Index (BMI) at screening is 18.5 or more but less than 25.0 kilogram per square metre (kg/m^2)
3. Written, informed consent to participate in the study based on the participant's own free will
4. Willing and able to comply with the requirements in the study after being fully informed of the requirements

Exclusion Criteria:

1. Male participants with reproductive potential who and whose partner do not agree to practice medically appropriate contraception (Note: throughout the study)
2. A history or complication of malignant tumor, lymphoma, leukemia, or lymphoproliferative disorder, a clinically significant disease requiring treatments within 8 weeks before the investigational product treatment, or a history of a clinically significant infection within 4 weeks before the investigational product treatment
3. With a psychiatric, digestive, hepatic, renal, respiratory, endocrine, hematologic, neural, or cardiovascular disease within 4 weeks before the investigational product treatment, a congenital metabolic abnormality, or otherwise a disease that may affect the drug assessments
4. With a surgical history (e.g., resection of the liver, kidney, or digestive tract, etc.) at screening that may affect the pharmacokinetics of the investigational product
5. Suspicion of having a clinically abnormal symptom or an organ impairment that requires treatments based on the history/complications at screening or physical findings, vital signs, electrocardiogram findings, or laboratory values at screening or baseline
6. Testing positive for human immunodeficiency virus (HIV) at screening
7. A positive response to a qualitative test for hepatitis B virus surface antigen (HBs antigen), hepatitis B virus core antigen (HBc) antibody, hepatitis C virus (HCV) antibody, or syphilis
8. Use of a prescription drug within 4 weeks before the investigational product treatment
9. Use of an over-the-counter drug within 2 weeks before the investigational product treatment
10. Receiving a vaccine within 4 weeks before the investigational product treatment
11. Ongoing participation in another clinical study or use of an investigational product or device within 16 weeks before the investigational product treatment while participating in another clinical study
12. Receiving blood transfusion within 12 weeks before the investigational product treatment, providing a whole-blood sample of 400 millilitre (mL) or more between 12 to 4 weeks before the investigational product treatment or a whole-blood sample of 200 mL or more within 4 weeks before the investigational product treatment, or giving blood components by pheresis within 2 weeks before the investigational product treatment

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Serum Concentrations of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
Change from Baseline in Serum Concentration of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
Peak Concentration (Cmax) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  Cmax is the maximum observed concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered.
Time to Peak Concentration (Tmax) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  Tmax is the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered.
Area Under the Concentration-time Curve (AUC 0-t) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  AUC 0-t is area under the concentration-time curve from time 0 to time of last quantifiable concentration for E3112.
Area Under the Concentration-time Curve (AUC∞) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  AUC∞ is area under the concentration-time curve from time 0 to infinity of E3112.
Half-life of Elimination (t1/2) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  t1/2 is the time required for the concentration of the drug to reach half of its original value.
Clearance (CL) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  CL is defined as the rate of drug elimination divided by the plasma concentration of the drug.
Volume of Distribution (Vd) of E3112 | Day 1: 0-24 hours; Day 8: 0-24 hours
  Vd is the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Day 1 to Day 43
Number of Participants with an Abnormal, Clinically Significant Hematology parameter value | Day 1 to Day 43
Number of Participants with an Abnormal, Clinically Significant Clinical Chemistry Parameter Value | Day 1 to Day 43
Number of Participants with an Abnormal, Clinically Significant Urine Value | Day 1 to Day 43
Number of Participants with Clinically Significant Change in Vital Signs | Day 1 to Day 43
Number of Participants with Clinically Significant Change in Electrocardiogram (ECG) | Day 1 to Day 43
Number of Participants with Clinically Significant Change in Physical Findings | Day 1 to Day 43
Number of Participants with Clinically Significant Change in Ophthalmological Findings | Day 1 to Day 43
Percentage of Participants with Serum Anti-E3112 Antibodies | Day 1 to Day 43

CONTACTS AND LOCATIONS:
Locations (1):
- EA Pharma Trial Site, Higashi, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No